CLINICAL TRIAL: NCT03343002
Title: Effect of Intravenous Fentanyl on the Occurrence of Postoperative Nausea and Vomiting According to Time of Administration Around the End of Tonsillectomy With or Without Adenoidectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 4-2017-0813
Record Dates: First submitted 2017-10-23; First posted 2017-11-17 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-08

CONDITIONS: Follicular Tonsillitis (Chronic)
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fentanyl at 10-15 min before end of surgery (Experimental)
  Interventions: Drug: fentanyl at 10-15 min before end of surgery
- fentanyl at end of surgery (Active Comparator)
  Interventions: Drug: fentanyl at end of surgery

INTERVENTIONS:
Drug: fentanyl at 10-15 min before end of surgery — Label 2 syringe is filled with 1mcg/kg of fentanyl, label 1 syringe is filled with same amount of saline solution. If the surgeon notifies the anesthesiologist 10-15 minutes before the end of the operation, the syringe drug labeled 1 will be administered intravenously(that is, normal saline ). At the end of the surgery, the syringe drug labeled 2 is administered intravenously((that is, 1mcg/kg of fentanyl)
  Arms: fentanyl at 10-15 min before end of surgery
Drug: fentanyl at end of surgery — Label 2 syringe is filled with 1mcg/kg of fentanyl, label 1 syringe is filled with same amount of saline solution. If the surgeon notifies the anesthesiologist 10-15 minutes before the end of the operation, the syringe drug labeled 1 will be administered intravenously(that is, normal saline ). At the end of the surgery, the syringe drug labeled 2 is administered intravenously((that is, 1mcg/kg of fentanyl)
  Arms: fentanyl at end of surgery

SUMMARY:
Fentanyl is a commonly used drug for the prevention of emergence agitation and reduction in postoperative pain in children receiving tonsillectomy. However, fentanyl can cause postoperative nausea and vomiting (PONV), which is a main target side effect that medical staff strives to prevent. However, recent meta-analysis showed that the incidence of PONV may be different depending on the time of administration of fentanyl. However, the research design of patients enrolled in each study, such as the age, the name of the operation, and the method of anesthesia, is not identical. The aim of this study was to evaluate the efficacy and safety of fentanyl in patients undergoing tonsillectomy with a prospective randomized controlled trial. Secondary outcomes include incidence and severity of emergence agitation and anesthesia recovery time, postanesthesia care unit (PACU) time, side effects.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients aged 3 to 7 years with ASA 1-II scheduled for tonsillectomy (or adenoidal tonsillectomy)

Exclusion Criteria:

* 1. History of developmental disorder, cognitive impairment, cerebral palsy
* 2. History of seizures(not simple febrile convulsions)
* 3. Upper respiratory infections
* 4. Structural airway disease predicting difficult airway
* 5. History of an adverse reaction, including allergic reactions to fentanyl

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 140 (Actual)
Dates: Start 2017-11-26 (Actual); Primary Completion 2018-08-27 (Actual); Study Completion 2018-08-27 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative nausea and vomiting | In 10-minute increments from immediately(less than 3 min) after entering PACU to departure
  Occurrence of nausea and vomiting- Described as yes/no (Observation of medical personnel or Subjective symptoms of the patient by the definition below) Nausea: "feeling of the urge to vomit" vomiting: "retching and any expulsion of liquid gastric contents"

SECONDARY OUTCOMES:
PAED scale score: *Pediatric Anesthesia Emergence Delirium scale: range 0-20 points. If the score is more than 12, it is considered to be EA occurrence. | In 10-minute increments from immediately(less than 3 min) after entering PACU to departure
  *Pediatric Anesthesia Emergence Delirium scale: range 0-20 points. If the score is more than 12, it is considered to be EA occurrence.
five-step EA scale: *five-step Emergence Agitation scale: range 1-5 score. If the score is 4 or more, it is regarded as EA occurrence. | In 10-minute increments from immediately(less than 3 min) after entering PACU to departure
  *five-step Emergence Agitation scale: range 1-5 score. If the score is 4 or more, it is regarded as EA occurrence.
FLACC score FLACC score (Face, Legs, Activity, Cry, Consolability scale): range 0-10. If the score is 4 or more, Pain control is considered necessary. | In 10-minute increments from immediately after entering PACU to departure
anesthesia recovery time | up to 1 day after end of surgery
  <1> time until regular respiration is possible after end of surgery , <2>time to extubate after end of surgery, and <3>eye opening time in response to initial verbal command after end of surgery
Occurrence of side effect | In 10-minute increments from immediately(less than 3 min) after entering PACU to departure
  airway obstruction, laryngospasm, desaturation, drowsiness, pruritus, hypotension, bradycardia

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No